CLINICAL TRIAL: NCT00066976
Title: Classification of Fetal Breathing Patterns in the Maturing Upper Airway: Spectral Waveform Analysis of Amniotic Fluid Flow Dynamics in Normal Development, Polyhydramnios, and Oligohydramnios
Brief Title: Studying Fetal Breathing Patterns
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030258; 03-CH-0258
Record Dates: First submitted 2003-08-07; First posted 2003-08-08 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-03-03

CONDITIONS: Pregnancy
Keywords: Prenatal; Respiration; Ultrasound; Prematurity; Diagnoses; Fetal Breathing-Movement; Doppler Sonography; Amniotic Fluid; Oligohydraminos; Polyhydraminos; Pregnancy
MeSH Terms: conditions — Respiratory Aspiration; Premature Birth; Disease

SUMMARY:
Some babies have difficulty breathing, sucking, and swallowing at birth. The purpose of this study is to determine (before birth) the variables that will predict whether a newborn will experience these problems.

Study participants will be pregnant women with a single fetus who are 18 years or older and who are scheduled to receive a standard prenatal ultrasound. Researchers will use the ultrasound to observe fetal motions associated with breathing, sucking, and swallowing on digital videotape. They will then review these tapes and take measurements that will help them document how breathing and swallowing develop.

DETAILED DESCRIPTION:
The aerodigestive tract is a complex system of integrated anatomical structures supporting ingestive and respiratory functions. The developmental origins of this system begin in utero where the prenatal growth of morphologic structures and their associated emerging behaviors form key physiologic foundations necessary to sustain life at birth. The quality of aerodigestive development is thus inextricably related to both the structural integrity of its growing anatomy and the emergence of processes that promote aerodigestive functioning. Our past research (NIH CC-00-99; NNMC #B99-089) focused specifically on emerging oropharyngeal, and laryngeal movements of neonatal swallowing and phonation. Through innovative sonographic techniques, this work documented ingestive development in the living fetus; however, respiratory aspects were not explored. Intuitively, disruptions to the fetal-maternal environment also influence respiratory development and, thus an arrest, disorder, or delay in maturation of upper airway mechanisms may directly affect subsequent postnatal respiratory function. Thus, the purposes of this protocol are to: 1) continue exploration of human fetal development by elucidating the association between upper airway growth and emerging prenatal respiratory function and, 2) determine identifiable patterns of normal respiratory maturation that may provide indicators of postnatal airway performance.

This initiative is based on the premise that amniotic fluid volumes are influenced by the integrity of upper airway mechanisms and thus are important for aerodigestive-related development and fetal well being. In a collaborative effort with National Naval Medical Center, this project will use a novel standardized 4-axis sonographic examination to quantify growth and respiratory-related fluid flow mechanics in the upper airway of the living human fetus. The use of this noninvasive ultrasound technique as part of the clinical prenatal examination will not only discriminate function at four upper airway sites (perinasal, oral, pharyngeal, and tracheal), but provide estimates of amniotic fluid flow volumes, inspiratory-expiratory fluid flow velocities and durations, and Doppler waveform patterns associated with fetal breathing and ingestive processes. This provides a method from which we can begin to explore how deviations in amniotic fluid regulation may be associated with morbidity and mortality and, the predictive utility of these indices in understanding conditions such as oligohydramnios or polyhydramnios. This germinal database will include healthy fetuses 16.0 to 39.6 weeks' gestational age and cases with polyhydramnios/oligohydramnios. By elucidating how developing structures integrate with emerging upper respiratory behaviors, this work will document the maturational events underlying normal function at birth that in turn may facilitate future clinical strategies for successful postnatal care.

ELIGIBILITY:
* INCLUSION CRITERIA:

Both normal controls and test cases will be openly recruited from referrals to the NNMC PAC.

Healthy mother's 18 years of age and over with uneventful, singleton pregnancies dated at 16.0 to 39.6 weeks gestation (based on last menstrual period) are the inclusion criteria.

EXCLUSION CRITERIA:

Mothers with pregnancies outside this dating and under 18 years of age are an exclusion factor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0
Dates: Start 2003-08-05; Study Completion 2008-03-03

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Naval Medical Center, San Diego, San Diego, California
  - National Naval Medical Center, Bethesda, Maryland

REFERENCES:
- [Background] Kliegman RM. Neonatal technology, perinatal survival, social consequences, and the perinatal paradox. Am J Public Health. 1995 Jul;85(7):909-13. doi: 10.2105/ajph.85.7.909. PMID 7604911